CLINICAL TRIAL: NCT05443737
Title: Evaluation of a Telehealth Oncofertility Care Intervention in Adolescent and Young Adult Cancer Patients: a Stepped Wedge Cluster Randomized Controlled Trial
Brief Title: Evaluation of a Telehealth Oncofertility Care Intervention in Adolescent and Young Adult Cancer Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Rady Children's Hospital, San Diego (Other); City of Hope Medical Center (Other)
Responsible Party: Principal Investigator, Hui-Chun Irene Su, Professor, University of California, San Diego
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 800780
Record Dates: First submitted 2022-06-24; First posted 2022-07-05 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Fertility Preservation
Keywords: Oncofertility; Fertility preservation; Adolescent and young adult cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized controlled trial
Who Masked: Care Provider
Masking Description: Fertility specialists and their support staff will be blinded to the intervention status of the cluster from which a patient is referred to minimize differences in counseling in patients whom they expect to receive financial navigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-component oncofertility care intervention (Experimental): Eligible cancer patients presenting to oncology clinical visits will receive care through the multi-component oncofertility care intervention.
  Interventions: Behavioral: Multi-component oncofertility care intervention
- Usual Care (No Intervention): Eligible cancer patients presenting to oncology clinical visits will receive usual care.

INTERVENTIONS:
Behavioral: Multi-component oncofertility care intervention — The multi-component oncofertility care intervention includes: (1) an adaptive and smart default electronic health record-based oncofertility needs screen and referral pathway, (2) telehealth oncofertility counseling as indicated, and (3) telehealth oncofertility financial navigation as indicated.
  Arms: Multi-component oncofertility care intervention

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a multi-component intervention to improve young cancer survivors' engagement in goal-concordant oncofertility care, concurrently with observing and gathering information on how the intervention is implemented. The investigators hypothesize that implementation of the intervention will result in increased young cancer survivors' engagement in goal-concordant oncofertility care.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed cancer or cancer relapse
* Primary language English or Spanish
* Receiving oncology care at participating clinical sites
* Ages 0 to 42 years if female
* Ages 0 to 50 years if male

Exclusion Criteria:

* Non-melanoma skin cancer, because primary treatment is excision with no infertility risk
* Metastatic/Stage IV non-thyroid solid tumors, because of poor prognosis

Ages: 0 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2800 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of reproductive-aged female and male patients (aged 12 to 39 years) who engage in goal-concordant oncofertility care | 12 weeks after oncology visit
  The proportion of eligible reproductive-aged male and female patients (aged 12 to 39 years) who engage in oncofertility services (1| an oncofertility needs screen, 2| referral to oncofertility consult, 3| oncofertility consult, and/or 4| fertility preservation services) that meet the patient's individual needs will be abstracted from medical records using standardized case report forms.
Decisional Conflict | 12 weeks after oncology visit
  The 16-item Decisional Conflict Scale (DCS) will be used to measure patients' decisional conflict for engaging in fertility preservation services. The DCS consists of 16 statements with 5 response options (ranging from strongly agree to strongly disagree) that measures the patient's perceptions of uncertainty in choosing options, feeling informed, values clarity, support in decision making, and effective decision making. The DCS total score will be dichotomized at 37.5 (scale 0-100; > 37.5 indicates high decisional conflict).

SECONDARY OUTCOMES:
Number of female (aged 0 to 42 years) and male (aged 0 to 50 years) patients who engage in goal-concordant oncofertility care | 12 weeks after oncology visit
  The proportion of eligible female and male patients (aged 0 to 42 years for females; 0 to 50 years for males) who engage in oncofertility services [1) an oncofertility needs screen, 2) referral to oncofertility consult, 3) oncofertility consult, and/or 4) fertility preservation services] that meet the patient's individual needs will be abstracted from medical records using standardized case report forms.
Number of female patients (aged 0 to 42 years) who engage in goal-concordant oncofertility care | 12 weeks after oncology visit
  The proportion of eligible female patients (aged 0 to 42 years) who engage in oncofertility services [1) an oncofertility needs screen, 2) referral to oncofertility consult, 3) oncofertility consult, and/or 4) fertility preservation services] that meet the patient's individual needs will be abstracted from medical records using standardized case report forms.
Number of male patients (aged 0 to 50 years) who engage in goal-concordant oncofertility care | 12 weeks after oncology visit
  The proportion of eligible male patients (aged 0 to 50 years) who engage in oncofertility services [1) an oncofertility needs screen, 2) referral to oncofertility consult, 3) oncofertility consult, and/or 4) fertility preservation services] that meet the patient's individual needs will be abstracted from medical records using standardized case report forms.

CONTACTS AND LOCATIONS:
Overall Officials: H. Irene Su, MD, MSCE, Principal Investigator — University of California, San Diego
Locations (4):
- United States (4):
  - City of Hope, Duarte, California
  - Cancer Resource Center of the Desert, El Centro, California
  - University of California San Diego, La Jolla, California
  - Rady Children's Hospital San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data generated during the study will be available from the principal investigator (H. Irene Su) upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication.
Access Criteria: Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to the principal investigator (H. Irene Su).

REFERENCES:
- [Derived] Romero SAD, Au L, Flores-Ortega RE, Helsten T, Palomino H, Kaiser BN, Echevarria M, Lukas K, Freeman K, Zou J, Aristizabal P, Armenian S, Su HI. Let's TOC Fertility: A stepped wedge cluster randomized controlled trial of the Telehealth Oncofertility Care (TOC) intervention in children, adolescent and young adult cancer survivors. Contemp Clin Trials. 2024 Jun;141:107537. doi: 10.1016/j.cct.2024.107537. Epub 2024 Apr 13. PMID 38614445